CLINICAL TRIAL: NCT00120653
Title: Metoclopramide to Treat Anemia in Patients With Myelodysplastic Syndrome (MDS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050201; 05-H-0201; NCT00238134 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2005-07-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Myelodysplastic Syndromes
Keywords: Reglan; Prolactin; MDS; Metoclopramide; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Metoclopramide

INTERVENTIONS:
Drug: Metoclopramide

SUMMARY:
This study will determine whether the medication metoclopramide can improve red blood counts in people who have myelodysplastic syndrome (MDS). MDS is thought to affect blood stem cells, which can result in low levels of red blood cells-that is, anemia-as well as low white blood cell and platelet counts. Patients with MDS are at risk for infection, spontaneous bleeding, and possible progression to leukemia, a cancer of bone marrow. Although bone marrow can produce some blood cells, this production can be decreased in patients with MDS. The definitive way to treat MDS is stem cell transplantation, but serious complications and a high risk of death make it unsuitable for patients older than age 60 or those who do not have a matched sibling donor. However, scientists have noted improvement in anemia by using metoclopramide, an inexpensive, commonly used medication that does not have many negative side effects. This study will evaluate the safety and effectiveness of that medicine for patients with MDS.

Patients ages 18 to 72 whose MDS would require low-intensity treatment-for example, with growth factor and transfusions-and who are not pregnant or breastfeeding may be eligible for this study. There will be about 60 participants.

Screening tests include a complete physical examination and medical history, during which patients will provide a list of current medications or supplements they are taking. There will be a collection of about 4 tablespoons of blood for analysis of blood counts as well as liver and kidney function. Patients may also undergo a magnetic resonance imaging (MRI) scan of their brain, but the procedure is optional. During the MRI, they will lie on a table that will slide into the enclosed tunnel of the scanner. The MRI takes about 20 to 30 minutes, and patients will be asked to lie as still as possible. There will also be a bone marrow biopsy, if patients have not had one done within 4 weeks of the start of this study. Eligible patients will take a 10 mg dose of metoclopramide by mouth, three times a day, for 20 weeks. They will be given a 4-week supply, which will be renewed monthly at each treatment visit. It is essential that patients be seen at NIH during the first, third, and fifth months of the study. Visits made in the meantime, at the second and fourth months, may be done at the office of their doctors who have referred them for the study, or at NIH. During the treatment visits, patients will be asked to update their medical history, health conditions, and use of medications or herbal supplements. There will also be a collection of about 1 tablespoon of blood for laboratory tests. Patients will be asked to make a similar follow-up visit 1 month after they stop taking metoclopramide, so that the response to treatment can be evaluated.

The use of metoclopramide may cause some people to feel dizzy, lightheaded, tired, or less alert than they are normally. For the first 24 to 48 hours, patients should be cautious when driving, using machinery, or performing hazardous activities. This medicine will add to the effects of alcohol and other central nervous system depressants-such as medicines for allergies and colds, tranquilizers, and prescription pain relievers. Patients need to check with the research team before taking any of those types of medicines, as well as herbal supplements, while using metoclopramide.

This study may or may not have a direct benefit for participants. For some, the drug may improve red blood cell counts and decrease the need for red cell transfusions. Knowledge gained in the study may help people in the future.

DETAILED DESCRIPTION:
Patients with myelodysplastic syndrome (MDS) present with low red blood cells, white blood cells and platelets, alone or in combination. The only definitive treatment is stem cell transplantation. Unfortunately, treatment-related mortality precludes the application of this procedure for most patients older than 60 years and those lacking a suitable matched sibling donor. A proportion of patients have been shown to respond to a wide variety of immunosuppressive agents, including cyclosporine (CSA) and antithymocyte globulin (ATG). However, nonresponse and relapse continue to be problematic. Therefore, most patients with MDS receive supportive treatment with transfusions and growth factors, such as erythropoietin (EPO) and G-CSF, to improve blood counts. However, growth factors are not always effective in improving cytopenias and iron overload is an inevitable long-term complication of red blood cell transfusions.

Recently, Abkowitz et al described clinically significant improvement in anemia in 3 of 9 patients with Diamond-Blackfan anemia (DBA) using metoclopramide, an inexpensive, commonly used medication with rare side effects. We hypothesize that therapy with metoclopramide might also benefit patients with other causes of refractory anemia, such as individuals with anemia due to MDS. We therefore propose this Phase II clinical trial to evaluate metoclopramide in the treatment of anemia in patients with MDS.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. MDS patients in IPSS risk group low or intermediate-1

     OR

     MDS patients in IPSS risk group intermediate-2 if greater than 60 years of age and not eligible for high intensity therapies, including intensive combination chemotherapy or hematopoietic cell transplant.
  2. Off all other treatments for MDS, except red blood cell transfusion support for at least 4 weeks.
  3. Anemia as defined by hemoglobin less than 11g/dL.
  4. Absolute reticulocyte count less than 60,000/microliter based on two baseline lab tests.
  5. Absolute neutrophil count greater than 200/microliter.
  6. Platelet count greater than 10,000/microliter.
  7. Ages 18 to 72.
  8. ECOG performance status less than or equal to 2.
  9. Ability to understand the investigational nature of the protocol and provide informed consent.

EXCLUSION CRITERIA:

1. MDS patients in high IPSS risk group.
2. Patients with secondary MDS.
3. Previous history of dystonic reaction and/or anaphylactic reaction to metoclopramide.
4. History of GI obstruction/perforation, pheochromocytoma, seizure disorders, creatinine clearance less than or equal to 50mL/min (estimated creatinine clearance = [weight (Kg) x (140-age) x (0.85 if female)]/[72 x (stable creatinine)], Parkinson's disease, breast cancer, clinically active depression, or hypertension due to pheochromocytoma
5. Current pregnancy (positive serum Beta-HCG if menstruating female), or unwilling to use a medically acceptable contraceptive or refrain from pregnancy if of childbearing potential
6. Concomitant drug therapy with high risks of extrapyramidal side effects (namely antipsychotic drugs including haloperidol, trifluoperazine, fluphenazine, thiothixene, perphenazine and pimozide).
7. Metoclopramide therapy 4 months prior to study enrollment.
8. Hyperprolactinemia prior to study implementation (prolactin greater than 200 ng/ml).

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07-14; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920